CLINICAL TRIAL: NCT06154759
Title: The Effect of Psycoeducation Based on The Watson's Human Caring Model Provided To The Relatives Of Palliative Care Patients on Hopelessness, Death Anxiıety, And Burden of Care
Brief Title: The Effect of Psychoeducation on Hopelessness, Death Anxiety and Caregiver Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Bilge Dilek Soyaslan, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.306565
Record Dates: First submitted 2023-06-21; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Support, Family
Keywords: Hopelessness; Death Anxiety; Burden of Care; Palliative care; Psychiatric Nursing
MeSH Terms: conditions — Necrophobia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The caregivers did not know which group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental caregiver group (Experimental): 33 of whom were in the experimental group and 33 in the control group, were included in the study. In the study, quantitative data were collected using Descriptive Characteristics Form, Beck Hopelessness Scale, Templer Death Anxiety Scale and Caregiver Strain Index, while qualitative data were collected using Structured Interview Form-1 and Structured Interview Form-2. Quantitative data collection tools were applied to the relatives of the patients in the experimental and control groups after the randomization group assignment within the scope of the pre-test. Psychoeducation was given to the relatives of the patients in the experimental group for 45-60 minutes once a week for eight weeks. Qualitative data were collected in sessions (sessions 2,3,5,7,8) and for this purpose, Structured Interview Form-1, Structured Interview Form-2, and audio recording were used. The same data collection tools were applied to the Experiment group for the post-test measurements after eight weeks.
  Interventions: Other: Watson Human Caring Model-based psychoeducation
- control caregiver group (No Intervention): In the study, quantitative data were collected using Descriptive Characteristics Form, Beck Hopelessness Scale, Templer Death Anxiety Scale and Caregiver Strain Index in control group. The control group received no intervention for eight weeks. The same data collection tools were applied to the Control group for the post-test measurements after eight weeks.

INTERVENTIONS:
Other: Watson Human Caring Model-based psychoeducation — It is a psychoeducation program based on the Watson human care model, one of the theories of the nursing profession, that includes healing processes, and consists of sessions that address the hopelessness, death anxiety and care burden of individuals.
  Arms: experimental caregiver group

SUMMARY:
This study was conducted to determine the effect of Watson Human Caring Model-based psychoeducation given to the relatives of patients receiving palliative care on hopelessness, death anxiety and the burden of care.

DETAILED DESCRIPTION:
This randomized controlled study was conducted with the relatives of patients hospitalized in the palliative care clinic of a training and research hospital in Ankara,Turkey. A total of 66 patient relatives, 33 of whom were in the experimental group and 33 in the control group, were included in the study. In the study, quantitative data were collected using Descriptive Characteristics Form, Beck Hopelessness Scale, Templer Death Anxiety Scale and Caregiver Strain Index, while qualitative data were collected using Structured Interview Form-1 and Structured Interview Form-2. Quantitative data collection tools were applied to the relatives of the patients in the experimental and control groups after the randomization group assignment within the scope of the pre-test. Then, individual psychoeducation was given to the relatives of the patients in the experimental group for 45-60 minutes once a week for eight weeks. Qualitative data were collected in these psychoeducation sessions (sessions 2,3,5,7,8) and for this purpose, Structured Interview Form-1, Structured Interview Form-2, and audio recording were used.

ELIGIBILITY:
Inclusion Criteria:

Ability to communicate in Turkish Ability to write in Turkish Being a primary relative of the patient The patient's relative has been in the clinic for at least one week in order to adapt to the caregiver role.

Does not have a visual, auditory or mental disability Only one relative of each patient participated in the study. Provide care by the patient's relatives for at least eight hours a day

Exclusion Criteria:

* Inability to speak Turkish
* Having a hearing impairment
* Lack of comprehension skills
* Participating in another psychoeducation program within the last year
* Having a physical or mental problem t

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Metting-Encounter | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  caregiver is informed about topics included in psychoeducation program and discussed in weekly.
  1. Beck Hopelessness Scale (BHS) was used to determine the hopelessness. The items are answered as "Yes-No". Total score is between 0-20. As the score of the scale increases; interpreted as an increase in hopelessness in individuals.
  2. Templer Death Anxiety (TDA)Scale was used to determine the death anxiety. The total score that can be obtained from the scale is between 0-15, and values of seven and above are interpreted as high death anxiety. The items are answered as "True-False".
  3. The Caregiver Strain Index (CSI)was used to determine care burden. The items in the scale are answered as "Yes-No". The total score of the scale is between 0-13,the average score of the scale is seven and above; interpreted as the burden of care in individuals.
  After psychoeducation,our aims are decreasing levels of
  1. For hopelessness, BHS used
  2. death anxiety, TDA used
  3. care burden, CSI used
Understanding palliative care | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Explaining the meaning of palliative care with the patient's relatives, discussing the common symptoms in patients.
  data from the qualitative stage; It was obtained by using structured interview forms of the relatives of the patients in the experimental group during psychoeducation program based on. In the 2nd, 3rd, 5th,7th sessions of psychoeducation, six questions were asked about the hopelessness, death anxiety and care burden. In this session, "What is the meaning of giving care to the relatives of the patients in the structured interview form-1? How did the caregiving process affect you?" A qualitative interview was conducted by asking the question.
Caregiving Process | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Meeting with the caregiver about the difficulties and gains of the caregiving process In this session, "Can you share your experiences about the difficulties of the caregiving process? Can you tell about your experiences that made you feel good during the caregiving process?" A qualitative interview was conducted by asking the question.
Hope- Sources of Hope | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Interviewing the caregiver about the importance of hope in life
Developing Hope | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Meeting with the patient's relatives about what can be done to improve hope. In this session, "Can you share your experiences about the concept of hope in the care process?", "You are here with your patient right now, you are helping him, what are your expectations for the next days?" A qualitative interview was conducted by asking the question.
Death- Death anxiety | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Interviewing the concept of death with the patient's relatives, providing information on what can be done to cope with death anxiety while caring for a patient with a terminal diagnosis.
Meaning of Life | It will be applied once a week for 45-60 minutes for up to 8 weeks.
  Interviewing with the caregiver about the meaning of life. In this session, "Can you share with me your end-of-life experiences in the caregiving process according to your culture and belief?" A qualitative interview was conducted by asking the question.
Last session | It will be applied once a week for 45-60 minutes for up to 8 weeks.Data collection forms (Descriptive Characteristics Form, Beck Hopelessness Scale, Templer Death Anxiety Scale and Caregiver Strain Index) applied again for post test to all caregivers.
  post test Beck Hopelessness Scale was used to determine the hopelessness levels of caregivers after psychoeducation. The scale has 20 items and these items are answered as "Yes-No". The total score is between 0-20. As the score of the scale increases; interpreted as an increase in hopelessness in individuals.
  Templer Death Anxiety Scale was used to determine the death anxiety of caregivers after psychoeducation The total score that can be obtained from the scale is between 0-15, and values of seven and above are interpreted as high death anxiety. The items in the scale are answered as "True-False".
  The Caregiver Strain Index was used to determine caregivers' burden of care after psychoeducation. items in the scale are answered as "Yes-No". The scale has no sub-dimensions. The scale's total score is between 0-13, and if the average score of the scale is seven and above; interpreted as the burden of care in individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge SOYASLAN, Master, Principal Investigator — Lecturer
Locations (1):
- Bilge Dilek SOYASLAN, Keçiören, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Best M, Leget C, Goodhead A, Paal P. An EAPC white paper on multi-disciplinary education for spiritual care in palliative care. BMC Palliat Care. 2020 Jan 15;19(1):9. doi: 10.1186/s12904-019-0508-4. PMID 31941486
- [Background] Valero-Cantero I, Casals C, Carrion-Velasco Y, Baron-Lopez FJ, Martinez-Valero FJ, Vazquez-Sanchez MA. The influence of symptom severity of palliative care patients on their family caregivers. BMC Palliat Care. 2022 Feb 28;21(1):27. doi: 10.1186/s12904-022-00918-3. PMID 35227246
- [Background] Del-Pino-Casado R, Priego-Cubero E, Lopez-Martinez C, Orgeta V. Subjective caregiver burden and anxiety in informal caregivers: A systematic review and meta-analysis. PLoS One. 2021 Mar 1;16(3):e0247143. doi: 10.1371/journal.pone.0247143. eCollection 2021. PMID 33647035
- [Background] Jors K, Seibel K, Bardenheuer H, Buchheidt D, Mayer-Steinacker R, Viehrig M, Xander C, Becker G. Education in End-of-Life Care: What Do Experienced Professionals Find Important? J Cancer Educ. 2016 Jun;31(2):272-8. doi: 10.1007/s13187-015-0811-6. PMID 25773135
- [Background] Alam S, Hannon B, Zimmermann C. Palliative Care for Family Caregivers. J Clin Oncol. 2020 Mar 20;38(9):926-936. doi: 10.1200/JCO.19.00018. Epub 2020 Feb 5. PMID 32023152
- [Background] Bischoff K, Yang E, Kojimoto G, Shepard Lopez N, Holland S, Calton B, Adkins SH, Cheng S, Miller BJ, Rabow MW. What We Do: Key Activities of an Outpatient Palliative Care Team at an Academic Cancer Center. J Palliat Med. 2018 Jul;21(7):999-1004. doi: 10.1089/jpm.2017.0441. Epub 2018 Feb 12. PMID 29431580
- [Background] Perpina-Galvan J, Orts-Beneito N, Fernandez-Alcantara M, Garcia-Sanjuan S, Garcia-Caro MP, Cabanero-Martinez MJ. Level of Burden and Health-Related Quality of Life in Caregivers of Palliative Care Patients. Int J Environ Res Public Health. 2019 Nov 29;16(23):4806. doi: 10.3390/ijerph16234806. PMID 31795461
- [Background] Nierop-van Baalen C, Grypdonck M, van Hecke A, Verhaeghe S. Associated factors of hope in cancer patients during treatment: A systematic literature review. J Adv Nurs. 2020 Jul;76(7):1520-1537. doi: 10.1111/jan.14344. Epub 2020 Mar 20. PMID 32133663
- [Background] Davis MP, Lagman R, Parala A, Patel C, Sanford T, Fielding F, Brumbaugh A, Gross J, Rao A, Majeed S, Shinde S, Rybicki LA. Hope, Symptoms, and Palliative Care. Am J Hosp Palliat Care. 2017 Apr;34(3):223-232. doi: 10.1177/1049909115627772. Epub 2016 Jul 10. PMID 26809826